CLINICAL TRIAL: NCT00714090
Title: Repetitive Transcranial Magnetic Stimulation Efficacy for Major Resistant Depression Compared or Associated With Venlafaxine : a Multicentric Study.
Brief Title: Repetitive Transcranial Magnetic Stimulation and Venlafaxine in Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Club rTMS et Psychiatrie (Other)
Collaborators: Ministry of Health, France (Other Government); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Dr Emmanuel POULET, Medical Doctor, Club rTMS et Psychiatrie
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAD-001
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Unipolar Depression
Keywords: repetitive Transcranial Magnetic Stimulation (rTMS); Major depressive disorders; Depression; Venlafaxine
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major; Depression | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator): Double active comparator : venlafaxine (150 mg/day) and rTMS (5 times/week)
  Interventions: Other: active venlafaxine and active rTMS-repetitive transcranial magnetic stimulator, Inomed and Alpine Biomed
- B (Experimental): active rTMS (5 times/week) and sham venlafaxine (150 mg/day)
  Interventions: Other: active rTMS -repetitive transcranial magnetic stimulator, Inomed and Alpine Biomed and sham venlafaxine
- C (Sham Comparator): sham rTMS (5 times/week) and active venlafaxine (150 mg/day)
  Interventions: Other: sham rTMS- repetitive transcranial magnetic stimulator, Inomed and Alpine Biomed and active venlafaxine

INTERVENTIONS:
Other: active venlafaxine and active rTMS-repetitive transcranial magnetic stimulator, Inomed and Alpine Biomed — active venlafaxine LP 75 mg : 1 capsule per day for 3 days, then 2 per day for 2 to 4 weeks, if necessary 3 per day the next 2 weeks.
  active rTMS : 5 sessions per week for 2 to 6 weeks
  Other Names: venlafaxine, Wyeth; repetitive transcranial magnetic stimulator, Inomed; repetitive transcranial magnetic stimulator, Alpine Biomed
  Arms: A
Other: active rTMS -repetitive transcranial magnetic stimulator, Inomed and Alpine Biomed and sham venlafaxine — active rTMS : 5 sessions per week for 2 to 6 weeks sham venlafaxine LP 75 mg : 1 capsule per day for 3 days, then 2 per day for 2 to 4 weeks, if necessary 3 per day the next 2 weeks.
  Other Names: repetitive transcranial magnetic stimulator, Inomed; repetitive transcranial magnetic stimulator, Alpine Biomed; venlafaxine, Wyeth
  Arms: B
Other: sham rTMS- repetitive transcranial magnetic stimulator, Inomed and Alpine Biomed and active venlafaxine — sham rTMS : 5 sessions per week for 2 to 6 weeks active venlafaxine LP 75 mg : 1 capsule per day for 3 days, then 2 per day for 2 to 4 weeks, if necessary 3 per day the next 2 weeks.
  Other Names: repetitive transcranial magnetic stimulator, Inomed; repetitive transcranial magnetic stimulator, Alpine Biomed; venlafaxine, Wyeth
  Arms: C

SUMMARY:
The purpose of this study is to assess the efficacy of add-on therapy with repetitive Transcranial Magnetic Stimulation (rTMS) and venlafaxine in the treatment of major depressive disorders compared to venlafaxine only (the optimal medication) and to rTMS only.

DETAILED DESCRIPTION:
rTMS parameters : Intensity of 120% of individually determined motor threshold; frequency : 1 Hz; 360 impulsions; on period : 1 min; off period : 30 s.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Clinical diagnosis of major depressive disorder (DSM-IV)
* HDRS-17 items > 20
* Failure of one antidepressant treatment (efficacious doses for 6 weeks at least)

Exclusion Criteria:

* I or II bipolar disorder
* Psychotic features
* Failure of one previous venlafaxine treatment
* Addiction comorbidity or schizophrenia comorbidity
* Involuntary hospitalization
* Seizures history
* Pregnancy or breastfeeding
* Somatic comorbidity able to impact on cognitive functions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2008-05; Primary Completion 2012-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is remission. It will be evaluated using the Hamilton Depression Rating Scale (HDRS-17 < 8)and Montgomery Asberg Depression Rating Scale (MADRS) | 2 to 6 weeks

SECONDARY OUTCOMES:
Onset of action for remission and response (HDRS-17 diminution > 50%) | 2 to 6 weeks
Anxiety will be assessed using the Covi Anxiety Scale. | 2 to 6 weeks
Side effects will be assessed using the UKU Scale. | 2 to 6 weeks
Evaluation of depression using 2 other scales : the Montgomery Asberg Depression Rating Scale (MADRS) and the Beck Depression Inventory scale (BDI-13) | 2 to 6 weeks
Onset of action using the Clinical Global Impressions scale (CGI) | 2 to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel POULET, MD, PhD, Principal Investigator — EA 4615 - SIPAD, Unité de Recherche UCB Lyon 1/CH Le Vinatier - Department of Psychiatry - Service du Pr d'AMATO
Locations (18):
- France (17):
  - C.H.U. Saint-Jacques - Service de Psychiatrie de l'Adulte, Besançon
  - C.H. Le Vinatier - EA 4166, UCB Lyon 1 - Department of Psychiatry - Service du Pr d'AMATO, Bron
  - C.H.U. Gabriel Montpied - Service de Psychiatrie et Psychologie Médicale - CMP A, Clermont-Ferrand
  - Hôpital Louis Mourier, Colombes
  - C.H.U. Dijon, Hôpital Général - Service de Psychiatrie et d'Addictologie, Dijon
  - C.H.U. de Grenoble, Hôpital sud - Département de Psychiatrie, Grenoble
  - ASM Limoux, Lézignan-Corbières
  - Hôpital Fontan - C.H.R.U. Lille, Lille
  - C.H. Sainte Marguerite, Marseille
  - CHU - Hôpital La Colombière, Montpellier
  - Hôpital Pasteur - CHU Nice, Nice
  - Hôpital Sainte Anne - Service Hospitalo-Universitaire de Santé Mentale et de Thérapeutique, Paris
  - C.H.U. de POITIERS, Poitiers
  - C.H.U. - C.H. Guillaume Régnier, Rennes
  - C.H.U. Charles Nicolle - Service Hospitalo-Universitaire de Psychiatrie, Rouen
  - EPS de Ville Evrard - Unité de Saint-Denis, Saint-Denis
  - CHU St Etienne - Hôpital Nord, Saint-Etienne
- Centre Hospitalier Princesse Grace, Monaco, Monaco

REFERENCES:
- [Derived] Brunelin J, Jalenques I, Trojak B, Attal J, Szekely D, Gay A, Januel D, Haffen E, Schott-Pethelaz AM, Brault C; STEP Group; Poulet E. The efficacy and safety of low frequency repetitive transcranial magnetic stimulation for treatment-resistant depression: the results from a large multicenter French RCT. Brain Stimul. 2014 Nov-Dec;7(6):855-63. doi: 10.1016/j.brs.2014.07.040. Epub 2014 Aug 7. PMID 25192980